CLINICAL TRIAL: NCT06858111
Title: Phase III Randomized Control Trial to Investigate the Safety and Efficacy of Fertilo Versus Medicult In Vitro Maturation (IVM)
Brief Title: Fertilo In Vitro Research Study and Trial
Acronym: FIRST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gameto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GAM-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: In Vitro Maturation of Oocytes
Keywords: IVF; IVM; In Vitro Fertilization; Fertilo; Gameto; infertility; fertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fertilo (Experimental): Immature cumulus-oocyte complexes (COCs) are oocytes surrounded by cumulus cells that have not yet matured. The COCs are cultured in Fertilo coculture condition then fertilized, grown to the blastocyst stage, vitrified, and later transferred for reproductive purpose.
  Interventions: Biological: Fertilo
- Medicult IVM® (Active Comparator): Immature COCs are cultured in the standard IVM system MediCult IVM® then fertilized, grown to the blastocyst stage, vitrified, and later transferred for reproductive purpose.
  Interventions: Device: Medicult IVM

INTERVENTIONS:
Biological: Fertilo — Fertilo is an engineered line of ovarian support cells that aid egg maturation.
  Arms: Fertilo
Device: Medicult IVM — MediCult IVM is a system of culture media designed for the in vitro maturation of immature oocytes.
  Arms: Medicult IVM®

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of using Fertilo for In vitro maturation (IVM) in participants 18-35 years of age. The main question it aims to answer is whether the use of Fertilo is superior to using Medicult IVM for In vitro maturation.

Researchers will compare the number of ongoing pregnancies at 12 weeks gestation for participants in each arm.

* Arm 1 participants will have all cumulus oocyte complexes (COCs), or eggs surrounded by helper cells, cultured in Fertilo for 30 hours.
* Arm 2 participants will have all cumulus oocyte complexes (COCs), or eggs surrounded by helper cells, cultured in Medicult IVM for 30 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Premenopausal, Age 18-35.
3. Body mass index (BMI) 21-40.
4. Candidate for IVF according to the ASRM definition (infertile for ≥12 months, require the use of donor sperm, or the inability to achieve a successful pregnancy based on a patient's medical, sexual, and reproductive history, age, physical findings, diagnostic testing, or any combination of those factors).
5. No contraindications to the use of oral contraceptive pills (OCP) or gonadotropins.
6. Plan to use embryos for transfer within 2 months of blastocyst cryopreservation.
7. Anti-mullerian hormone (AMH) ≥ 3 ng/mL within 6 months of Screening/Visit 1 or assessed at the screening visit.
8. Normal uterine cavity as assessed by hysteroscopy, hysterosalpingography or sonohysterography within 12 months of Screening/Visit 1 or assessed at the screening visit.
9. Having adequate visualization of both ovaries, without evidence of significant abnormality/pathology or major cyst documented by transvaginal ultrasound within 3 months of screening or assessed during screening period.
10. No endometriosis of American Fertility Society (AFS) grade 3 or 4 or presence of endometrioma.
11. Minimum of 1 month without treatment with either clomiphene citrate, GnRH agonist or gonadotropins prior to start of ovarian stimulation.
12. Have a male partner with semen analysis within the past 12 months prior to randomization considered adequate to proceed with intracytoplasmic sperm injection (ICSI) according to the center's standard practice. If this criterion is not met, the subject can only be entered if donor sperm will be used.

Exclusion Criteria:

1. History of recurrent pregnancy loss (defined as >2 clinical pregnancies without live birth).
2. Baseline prolactin levels greater than 30 ng/ml
3. Male: requirement for retrograde ejaculation procedures or surgical sperm retrievals.
4. Any clinically relevant pathology that in the judgment of the investigator could impair embryo implantation or pregnancy continuation.
5. Use of preimplantation genetic testing (PGT) of oocytes, embryos, or transferred blastocysts during participation in the study.
6. Use of donated oocytes, embryos or blastocysts for this treatment cycle while participating in the study or use of oocytes, embryos, or blastocysts from a previous treatment cycle.
7. Participation in a concurrent clinical trial or in another investigational drug trial within the past 2 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender females, non-binary females of childbearing potential
Enrollment: 500 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Demonstration of the superiority of Fertilo compared to the currently approved MediCult IVM® for infertility treatment via IVF procedures. | 12 weeks gestation
  Cumulative ongoing pregnancy from cycles initiated within 6 months post-randomization. The primary endpoint of ongoing pregnancy is assessed at 12 weeks gestation or later. Cumulative ongoing pregnancy is determined using the cumulative outcome of up to the first two embryo transfers. Subjects with a detectable fetal heartbeat, considered normal and healthy, are considered as having achieved an ongoing pregnancy. "Normal" will be determined as expected for the gestational age ranging from 110 bpm to 180 bpm and measured via ultrasound. Ongoing pregnancy is recorded as either a Yes or No for normal fetal heart rate present for each of the Subject's transfer cycles. Subjects without an ongoing pregnancy assessment are considered as a No unless a later observation indicates otherwise (i.e., a live birth). Cumulative ongoing pregnancy is derived as either a Yes, if at least one of the first two embryo transfers achieves an ongoing pregnancy, or a No otherwise.

SECONDARY OUTCOMES:
Metaphase II (MII) Formation | 30 hours post-oocyte retrieval
  MII formation rate is assessed at 30 hours post-oocyte retrieval. A Metaphase II (MII) oocyte is defined as an oocyte with a first polar body (PB1). The MII formation rate is measured as a Subject's total number of MII oocytes divided by their total number of COCs. The MII formation rate is multiplied by 100 and expressed as a percentage.
Fertilization Rate | 16-18 hours post-ICSI
  Fertilization rate is assessed at 16-18 hours post-ICSI. Fertilized embryos displaying 2 pronuclei and 2 polar bodies are considered normally fertilized. Fertilized embryos with no pronuclei are considered not fertilized. Fertilized embryos with one pronuclei are held to determine cleavage, as pronuclei visualization timing may mask the second pronucleus. The fertilization rate is measured as a Subject's total number of fertilized embryos divided by their total number of COCs. The fertilization rate is multiplied by 100 and expressed as a percentage.
Embryo cleavage rate | Day 3 post-ICSI
  Embryo cleavage rate is assessed at day 3 post-ICSI. Embryos with 2 or more cells are considered as cleaved. Fertilized embryos displaying a single cell will be considered not cleaved. The cell cleavage rate is measured as a Subject's total number of embryos considered as cleaved divided by their total number of COCs. The cell cleavage rate is multiplied by 100 and expressed as a percentage.
High quality blastocyst formation rate. | Day 5, 6, and 7 post-ICSI
  High quality blastocyst formation rate is assessed at day 5, 6 and 7 post-ICSI. Embryos that have successfully passed the morula stage, as indicated by cavitation, will be designated as blastocysts and will be graded according to the Gardner Scale. Blastocysts having a Gardner Scale score of 3CC or higher are considered as high quality blastocysts. The high quality blastocyst formation rate is measured as a Subject's total number of high quality blastocysts divided by their total number of COCs. The high quality blastocyst formation rate is multiplied by 100 and expressed as a percentage.
High quality vitrified blastocyst rate. | Day 5, 6, and 7 post-ICSI
  High quality vitrified blastocyst rate is assessed at day 5, 6 and 7 post-ICSI. Embryos deemed high quality, as measured by a Gardner score of 3CC of greater, that have been vitrified, a method of rapid cryopreservation for future embryo transfer, will be designated as high quality vitrified blastocysts. The high quality vitrified blastocyst rate is measured as a Subject's total number of high quality blastocysts that are vitrified divided by their total number of COCs. The high quality vitrified blastocyst rate is multiplied by 100 and expressed as a percentage.
Cumulative biochemical pregnancy. | 10 to 14 days following FET
  Cumulative biochemical pregnancy from cycles initiated within 6 months post randomization. Biochemical pregnancy is assessed at 10 to 14 days following FET. Cumulative biochemical pregnancy is determined using the cumulative outcome of up to the first two embryo transfers. Subjects with BHCG value greater than 5 mIU/mL on two separate tests are considered as achieving biochemical pregnancy. Biochemical pregnancy is recorded as either a Yes or No for each of the Subject's transfer cycles. Subjects without a biochemical pregnancy assessment are considered as a No unless a later observation indicates otherwise (i.e., a clinical pregnancy, ongoing pregnancy, or live birth). Cumulative biochemical pregnancy is derived as either a Yes, if at least one of the first two embryo transfers achieves a biochemical pregnancy, or a No otherwise.
Cumulative clinical pregnancy. | 4-6 weeks gestation
  Cumulative clinical pregnancy from cycles initiated within 6 months post randomization is assessed at 4-6 weeks gestation. Cumulative clinical pregnancy is determined using the cumulative outcome of up to the first two embryo transfers. Subjects with a gestational sac visualized with TVU are considered as having achieved a clinical pregnancy. Clinical pregnancy is recorded as either a Yes or No for each of the Subject's transfer cycles. Subjects without a clinical pregnancy assessment are considered as a No unless a later observation indicates otherwise (i.e., an ongoing pregnancy or live birth). Cumulative clinical pregnancy is derived as either a Yes, if at least one of the first two embryo transfers achieves a clinical pregnancy, or a No otherwise.
Cumulative live birth. | Greater than 24 weeks gestation
  Cumulative live birth from cycles initiated within 6 months post-randomization. Live birth is confirmed at >24 weeks gestation by the presence of signs of life such as breathing, heartbeat, pulsation of the umbilical cord, or definitive movement of voluntary muscles. Cumulative live birth is determined using the cumulative outcome of up to the first two embryo transfers. Subjects with at least one neonate meeting the definition of live birth are considered as having achieved a live birth. Live birth is recorded as either a Yes or No for each of the Subject's transfer cycles. Subjects without a live birth assessment are considered as a No. Cumulative live birth is derived as either a Yes, if at least one of the first two embryo transfers achieves a live birth, or a No otherwise.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - HRC Fertility, Encino, California
  - Florida Fertility Institute, Clearwater, Florida
  - IVF Florida, Pembroke Pines, Florida
  - Shady Grove Fertility, Rockville, Maryland
  - Columbia University Fertility Center, New York, New York
  - Reach Fertility, Charlotte, North Carolina
  - Conceptions Fertility, Raleigh, North Carolina
  - Care Fertility, Bedford, Texas
  - Dallas Fort Worth Fertility Associates, Dallas, Texas
  - Shady Grove Houston, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Requestord will need to contact clinicaltrials@gametogen.com and sign a data access agreement.